CLINICAL TRIAL: NCT05752799
Title: Evaluation of the Stress Response in Bariatric Surgery With and Without the Use of Opioids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: G.Gennimatas General Hospital (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Panagiotis Chatzistavridis, Principal Investigator, G.Gennimatas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 31235/1.12.2022
Record Dates: First submitted 2023-02-11; First posted 2023-03-03 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Opioid Use, Unspecified; Bariatric Surgery Candidate
Keywords: morbid obesity; opioid free anaesthesia; nociception level; analgesia; bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Infusions will be prepared by independent staff not involved in the study. All preparations will be alike in the volume and appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid Based Anaesthesia (Active Comparator): This arm will receive:
  * 2 mcg/kg fentanyl in 10 ml volume
  * 0.2 mL/kg/h remifentanil infusion
  * 0.1 mg/kg morphine
  Interventions: Drug: Opioid based anesthesia
- Opioid Free Anaesthesia (Active Comparator): This arm will receive
  * 40 mg/kg magnesium sulfate in 100 ml N/S infusion
  * 0.4 mcg/kg dexmedetomidine, max total dose 50mcg in 50 ml N/S infusion
  * 0.3 mg/kg ketamine in 10 ml volume
  * 0.2 ml/kg of the Multimix regimen in 100 ml N/S infusion as a bolus (The Multimix regimen consists of 50mcg dexmedetomidine, 500 mg lidocaine and 50mg ketamine).
  * 0.2 ml/kg/h of the Multimix regimen in 100 ml N/S infusion as a continuous infusion
  Interventions: Drug: Opioid Free Anaesthesia

INTERVENTIONS:
Drug: Opioid Free Anaesthesia — * 40 mg/kg magnesium sulfate in 100 ml N/S infusion
  * 0.4 mcg/kg dexmedetomidine, max total dose 50mcg in 50 ml N/S infusion
  * 0.3 mg/kg ketamine in 10 ml volume
  * 0.2 ml/kg of the Multimix regimen in 100 ml N/S infusion as a bolus (The Multimix regimen consists of 50mcg dexmedetomidine, 500 mg lidocaine and 50mg ketamine).
  * 0.2 ml/kg/h of the Multimix regimen in 100 ml N/S infusion as a continuous infusion. Except for standard analgesic strategies, both groups will receive fentanyl as a rescue dose (1mcg/kg) based on a nociceptive level value > 25 or elevation of Heart Rate and/or Blood Pressure >20%.
  Placebo infusions of normal saline will be prepared to enable blinding.
  Arms: Opioid Free Anaesthesia
Drug: Opioid based anesthesia — * 2 mcg/kg fentanyl in 10 ml volume
  * 0.2 mL/kg/h remifentanil infusion
  * 0.1 mg/kg morphine. Except for standard analgesic strategies, both groups will receive fentanyl as a rescue dose (1mcg/kg) based on a nociceptive level value > 25 or elevation of Heart Rate and/or Blood Pressure >20%.
  Placebo infusions of normal saline will be prepared to enable blinding.
  Arms: Opioid Based Anaesthesia

SUMMARY:
The goal of this clinical trial is to compare Opioid Free and Opioid Based Anaesthesia in patients undergoing sleeve gastrectomy. The main questions it aims to answer are:

* Will the total dose of intraoperative opioid be reduced?
* Will there be difference in pain scores between groups? Participants will be managed with the Nociceptive Level Index algorithm to guide intraoperative analgesia.

The Opioid Free Anaesthesia Group will be administered the Multimix infusion (Magnesium sulfate, dexmedetomidine, ketamine). The Opioid Based Anaesthesia Group will receive fentanyl as a bolus dose and remifentanil infusion.

Rescue fentanyl bolused will be injected as appropriate according to nociceptive level (NOL) values.

DETAILED DESCRIPTION:
Opioid Free Anaesthesia has attracted the attention of clinicians since the outbreak of the opioid pandemic in the USA. It has been correlated with less intraoperative and postoperative opioid use. The Nociceptive Level Index algorithm allows for intraoperative monitoring of the nociceptive pathways and targeted pain management. Furthermore, it is known that morbidly obese patients may benefit from opioid sparing techniques.

Our aim is to investigate the effect of Opioid Free versus Opioid Based Anesthesia on postoperative pain in patients undergoing sleeve gastrectomy.

In this randomized, double blind clinical trial, patients will be allocated into two groups based on intraoperative pain management. Apart from recording postoperative pain scores, blood samples will be collected intraoperatively to evaluate the stress response among the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age >18y and <75y
* morbid obesity confirmed diagnosis
* American Society of Anesthesiologists (ASA) II-III
* elective laparoscopic sleeve gastrectomy surgery
* signed informed consent

Exclusion Criteria:

* bradycardia, bundle branch block, hypotension, postural hypotension
* obstructive sleep apnoea
* history of depression
* chronic corticosteroid use or intraoperative administration of more than 8mg of prednisolone or equivalent
* refusal to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Visual Analogue Scale (VAS) score | 6 hours after surgery
  The patient will be interviewed regarding postoperative pain using Visual Analogue Scale, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable

SECONDARY OUTCOMES:
First demand for supplementary analgesia | Up to 24 hours postoperatively
  The time to the first demand for supplementary analgesia will be recorded for every patient enrolled.
Postoperative VAS score | 24 hours
  The patient will be interviewed regarding postoperative pain using Visual Analogue Scale, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable
Perioperative trend of Adrenaline | At baseline, at the end of the operation, 24 hours after surgery
  Blood will be collected to measure the plasma adrenaline levels
Perioperative trend of Noradrenaline | At baseline, at the end of the operation, 24 hours after surgery
  Blood will be collected to measure the plasma Noradrenaline levels
Perioperative trend of Cortisol | At baseline, at the end of the operation, 24 hours after surgery
  Blood will be collected to measure the plasma Cortisol levels
Perioperative trend of Dopamine | At baseline, at the end of the operation, 24 hours after surgery
  Blood will be collected to measure the plasma Dopamine levels

CONTACTS AND LOCATIONS:
Locations (1):
- G.Gennimatas General Hospital, Athens, Greece

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT05752799/Prot_SAP_000.pdf